CLINICAL TRIAL: NCT05648708
Title: Comparing Combined Adductor Canal & Sciatic Nerve Block and Femoral & Sciatic Nerve Block for Postoperative Analgesia in Patients Undergoing Total Knee Replacement Surgery; A Prospective, Randomized, Controlled Study
Brief Title: Combined Adductor&Sciatic Nerve Block vs Femoral&Sciatic Nerve Block in Total Knee Replacement Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Responsible Party: Principal Investigator, Gokhan Sertcakacilar, MD, Principal investigator, Bakirkoy Dr. Sadi Konuk Research and Training Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: 2022-361
Record Dates: First submitted 2022-11-28; First posted 2022-12-13 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Orthopedic Disorder; Total Knee Replacement; Post Operative Pain; Surgery
Keywords: Femoral Nerve Block; Sciatic Nerve Block; Adductor Canal Block; General anesthesia; Orthopedic surgery; Post Operative Analgesia
MeSH Terms: conditions — Musculoskeletal Diseases; Pain, Postoperative | interventions — Bupivacaine; Prilocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group AS (Active Comparator): The investigators will perform an adductor canal block and sciatic nerve block on that patient group for postoperative analgesia
  Interventions: Procedure: Combine Adductor Canal & Sciatic Nerve Block; Drug: Bupivacaine and prilocaine hydrochloride
- Group FS (Active Comparator): The investigators will perform femoral and sciatic nerve blocks on that patient group for postoperative analgesia
  Interventions: Procedure: Combine Femoral & Sciatic Nerve Block; Drug: Bupivacaine and prilocaine hydrochloride

INTERVENTIONS:
Procedure: Combine Adductor Canal & Sciatic Nerve Block — The investigators will perform a combined adductor canal & sciatic nerve block on that patient group for postoperative analgesia
  Arms: Group AS
Procedure: Combine Femoral & Sciatic Nerve Block — The investigators will perform a combined femoral & sciatic nerve block on that patient group for postoperative analgesia
  Arms: Group FS
Drug: Bupivacaine and prilocaine hydrochloride — The investigators will perform a combined adductor canal & sciatic nerve block on that patient group for postoperative analgesia with bupivacaine and prilocaine hydrochloride
  Arms: Group AS
Drug: Bupivacaine and prilocaine hydrochloride — The investigators will perform a combined femoral & sciatic nerve block on that patient group for postoperative analgesia with bupivacaine and prilocaine hydrochloride
  Arms: Group FS

SUMMARY:
Knee joints, one of the largest and most functional joints of the human body, have great features to provide ideal body posture and movement. In patients with knee osteoarthritis in whom pain and functional loss continue to increase despite conservative and medical burden, they are evaluated by orthopedic surgeons for surgical treatment. Total knee replacement (TKR) surgery is aimed to eliminate the existing pain, restore and carry the movements, to protect the characteristics of the deformities and the quality of life.

Pain can be very severe after TKR surgery, which is very common in the middle and elderly patient population today. In the postoperative period, untreated pain prevents early physical therapy practices and restricts postoperative knee rehabilitation and recovery, but it also has negative effects on the respiratory, gastrointestinal, renal, and central nervous systems. Effective management of postoperative acute pain can reduce these complications and the risk of developing chronic pain.

In this study, investigators hypothesized that combined adductor canal and sciatic nerve block, applied with postoperative ultrasound guidance to patients who will undergo TKR surgery under general anesthesia, will provide effective analgesia, less opioid consumption, and faster ambulation time, similar to combined femoral and sciatic nerve block.

DETAILED DESCRIPTION:
As a result of the power analysis investigators conducted for this study, the minimum sample size was calculated as 34 people for each group, 68 people in total, at the 95% confidence interval.

68 patients who meet the inclusion criteria will be included in our study. Patients will be randomized and divided into 2 groups. Accordingly, femoral and sciatic nerve blocks will be applied to 34 patients, and adductor canal and sciatic nerve blocks will be applied to 34 patients.

ELIGIBILITY:
Inclusion Criteria:

* Ages of 40-85
* ASA I-III
* Patients who will undergo total knee replacement surgery under general anesthesia

Exclusion Criteria:

* Patients with deformity and pathology in the thigh region
* Clinically known local anesthetic allergy
* Clinically diagnosis of opioid, alcohol and substance dependence
* Patients who cannot perceive and evaluate pain such as psychiatric illness, mental retardation, dementia
* Morbid obesity (body mass index> 40 kg m2)

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2022-11-14 (Actual); Primary Completion 2023-08-21 (Actual); Study Completion 2023-10-23 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure of the study is the patients' postoperative pain scores (NRS) | 72 hours postoperatively
  Numerical rating scale (NRS) at 1, 6, 12, 18, 24, 48, 72th hours. NRS assessment score ranges from 0-10. 0 = no pain 10 = worst pain imaginable

SECONDARY OUTCOMES:
The secondary outcome measure will be total opioid consumption in the first 72 hours postoperatively | Three days postoperatively
  PCA device will be prepared with 4 mg tramadol (400 mg/100 cc) per ml and total opioid consumption for 72 hours will be noted

OTHER OUTCOMES:
Side effects due to postoperative opioid consumption, rescue analgesic requirements, hemodynamic parameters and satisfaction with analgesic method | Three days postoperatively
  Opioid side effects ( Nausea, Vomiting, Constipation, Itching, Mental cloudiness, Sweating, Fatigue, Drowsiness ) will be evaluated and noted as none-mild-moderate-severe for 72 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Bakirkoy Dr. Sadi Konuk Research and Training Hospital, Istanbul, Bakirkoy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Data available from the publication date can start. NRS scores and Opioid consumption and side effects will be shared. If requested, data will be shared with anesthesiologists dealing with postoperative analgesia in patients undergoing total knee replacement surgery
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Two year within the publication date.

REFERENCES:
- [Background] Auroy Y, Narchi P, Messiah A, Litt L, Rouvier B, Samii K. Serious complications related to regional anesthesia: results of a prospective survey in France. Anesthesiology. 1997 Sep;87(3):479-86. doi: 10.1097/00000542-199709000-00005. PMID 9316950
- [Background] Sladjana UZ, Ivan JD, Bratislav SD. Microanatomical structure of the human sciatic nerve. Surg Radiol Anat. 2008 Nov;30(8):619-26. doi: 10.1007/s00276-008-0386-6. Epub 2008 Jul 23. PMID 18648720
- [Background] Currin SS, Mirjalili SA, Meikle G, Stringer MD. Revisiting the surface anatomy of the sciatic nerve in the gluteal region. Clin Anat. 2015 Jan;28(1):144-9. doi: 10.1002/ca.22449. Epub 2014 Aug 8. PMID 25131147
- [Background] Bozkurt M, Yilmazlar A, Bilgen OF. [Comparing the effects of analgesia techniques with controlled intravenous and epidural on postoperative pain and knee rehabilitation after total knee arthroplasty]. Eklem Hastalik Cerrahisi. 2009;20(2):64-70. Turkish. PMID 19619108
- [Background] Gray AT, Collins AB. Ultrasound-guided saphenous nerve block. Reg Anesth Pain Med. 2003 Mar-Apr;28(2):148; author reply 148. doi: 10.1053/rapm.2003.50000. No abstract available. PMID 12677627